CLINICAL TRIAL: NCT01983969
Title: Azacitidine/Vorinostat/GemBuMel With Autologous Stem-Cell Transplant (SCT) in Patients With Refractory Lymphomas
Brief Title: Aza-SAHA-GBM With AutoSCT for Refractory Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0186; NCI-2014-01025 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Cancers; Lymphoma
Keywords: Advanced Cancers; Lymphoma; Recurrent Hodgkin's; non-Hodgkin's lymphoma; Stem cell transplant; Azacitidine; 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine; Vorinostat; SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza; Gemcitabine; Gemcitabine Hydrochloride; Gemzar; Busulfan; Busulfex; Myleran; Melphalan; Alkeran; Dexamethasone; Decadron; Caphosol; Glutamine; Enterex; Glutapak-10; NutreStore; Resource; GlutaSolve; Sympt-X G.I.; Sympt-X; Pyridoxine; Rituximab; Rituxan
MeSH Terms: conditions — Lymphoma; Lymphoma, Non-Hodgkin | interventions — Azacitidine; Vorinostat; Gemcitabine; Busulfan; Melphalan; Dexamethasone; Calcium Dobesilate; Glutamine; Health Resources; Pyridoxine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Azacitidine + Vorinostat + Gemcitabine + Busulfan + Melphalan (Experimental): Busulfan test dose 32 mg/m2 by vein either as outpatient before Day -12 or as inpatient on Day -11. Busulfan pharmacokinetics performed with test dose and first dose on Day -8. Doses on Days -6 and -5 adjusted to target an AUC of 4,000 microMol.min-1. Dexamethasone 8 mg by vein twice a day from Day -11 AM to Day -2 PM. Caphosol oral rinses 30 mL four times a day used from Day -9. Oral glutamine, 15 g four times a day, swished, gargled and swallowed from Day -9. Pyridoxine 100 mg by vein or mouth three times a day from Day -1. Vorinostat 1000 mg by vein on Day -11 through Day -2. Gemcitabine loading dose 75 mg/m2 by vein followed by 22775 mg/m2 by vein on Day -8. Melphalan 60 mg/m2 by vein on Days -3 and -2. Azacitidine starting dose 15 mg/ m2 by vein on Day -11. Stem cell transplant on Day 0. Patients with CD20+ tumors receive rituximab 375 mg/m2 by vein on Days -9.
  Interventions: Drug: Azacitidine; Drug: Vorinostat; Drug: Gemcitabine; Drug: Busulfan; Drug: Melphalan; Drug: Dexamethasone; Other: Caphosol; Drug: Glutamine; Drug: Pyridoxine; Drug: Rituximab

INTERVENTIONS:
Drug: Azacitidine — Starting dose 15 mg/ m2 by vein on Day -11.
  Other Names: 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
Drug: Vorinostat — 1000 mg by vein on Day -11 through Day -2.
  Other Names: SAHA; Suberoylanilide Hydroxamic Acid; MSK-390; Zolinza
Drug: Gemcitabine — Loading dose 75 mg/m2 by vein followed by 22775 mg/m2 by vein on Day -8.
  Other Names: Gemcitabine Hydrochloride; Gemzar
Drug: Busulfan — Busulfan test dose 32 mg/m2 by vein either as outpatient before Day -12 or as inpatient on Day -11. Busulfan pharmacokinetics performed with test dose and first dose on Day -8. Doses on Days -6 and -5 adjusted to target an AUC of 4,000 microMol.min-1.
  Other Names: Busulfex; Myleran
Drug: Melphalan — 60 mg/m2 by vein on Days -3 and -2.
  Other Names: Alkeran
Drug: Dexamethasone — 8 mg by vein twice a day from Day -11 AM to Day -2 PM.
  Other Names: Decadron
Other: Caphosol — Caphosol oral rinses 30 mL four times a day used from Day -9.
Drug: Glutamine — Oral glutamine, 15 g four times a day, swished, gargled and swallowed from Day -9.
  Other Names: Enterex; Glutapak-10; NutreStore; Resource; GlutaSolve; Sympt-X G.I.; Sympt-X
Drug: Pyridoxine — 100 mg by vein or mouth three times a day from Day -1.
Drug: Rituximab — 375 mg/m2 by vein on Days -9.
  Other Names: Rituxan

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of azacitidine that can be given with vorinostat, gemcitabine, busulfan, and melphalan, with a stem cell transplant, and with or without rituximab. Researchers also want to learn about the safety and level of effectiveness of this combination.

DETAILED DESCRIPTION:
Study Groups:

If you have been found to be eligible to take part in this study and you agree, you will be assigned to a dose level of azacitidine based on when you join this study. Up to 7 dose levels of azacitidine will be tested. At least 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of azacitidine is found.

All participants will receive the same dose level of vorinostat, gemcitabine, busulfan, and melphalan, and all patients with B-cell cancer will receive the same dose of rituximab. However, if the first group has bad side effects, the dose level of gemcitabine may be lowered for all other groups.

Busulfan Test Dose:

You will receive a test dose of busulfan by vein over about 60 minutes. This low-level test dose of busulfan is to check how the level of busulfan in your blood levels changes over time. This information will be used to decide the next dose needed to reach the target blood level that matches your body size. You will most likely receive this as an outpatient during the week before you are admitted to the hospital. If it cannot be given as an outpatient, you will be admitted to the hospital on Day -12 (12 days before your stem cells are returned to your body) and the test dose will be given on Day -11.

About 11 samples of blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing of busulfan. PK testing measures the amount of study drug in the body at different time points and will help the study doctor determine what your dose of busulfan should be on study. These blood samples will be drawn at various timepoints before you receive busulfan and over about the next 11 hours. The blood samples will be repeated again on the first day of high-dose busulfan treatment (Day -8). A temporary heparin lock line will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed for technical or scheduling reasons, you will receive the standard fixed dose of busulfan.

On Days -14, -13, and -12, you will receive palifermin by vein over about 30 seconds each day to help decrease the risk of side effects in the mouth and throat.

Study Drug Administration (for all patients):

In stem cell transplants, the days before you receive your stem cells are called minus days. The day you receive the stem cells is called Day 0. The days after you receive your stem cells are called plus days.

Beginning on Day -9, you will swish the liquids caphosol and glutamine in your mouth 4 times a day, for about 2 minutes each time. You will swish these liquids every day until you leave the hospital. You will swallow the glutamine. These drugs are used to help decrease the risk of side effects in the mouth and throat.

On Day -11 through Day -2, you will take vorinostat by mouth, with food. One hour later each day, you will receive azacitidine by vein over 1 hour. You will receive dexamethasone by vein 2 times each day.

If you have a B-cell cancer, you will receive rituximab (a treatment used for certain lymphomas) by vein over 3-6 hours as part of standard of care, on Day -9.

On Day -8, you will receive gemcitabine by vein over 4 ½ hours.

On Days -8, -7, -6, and -5, you will receive busulfan by vein over 2 hours.

On Day -3, you will receive gemcitabine by vein over 4 ½ hours and then melphalan by vein over 30 minutes.

On Day -2, you will receive melphalan by vein over 30 minutes.

On Day -1, you will rest (you will not receive chemotherapy).

On Day 0, you will receive your stem cells by vein over about 30-60 minutes.

You will receive 3 more doses of palifermin by vein over 15-30 seconds on Days 0, +1, and +2.

As part of standard care, you will receive G-CSF (filgrastim) as an injection just under your skin 1 time each day starting on Day +5 until your blood cell levels return to normal.

Study Tests:

About 100 days after the transplant:

* You will have a physical exam.
* Blood (about 4 teaspoons) and urine will be collected for routine tests.
* If the doctor thinks it is needed, you may have a bone marrow aspiration and biopsy to check the status of the disease. To collect a bone marrow aspiration/biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.

Length of Study:

As part of standard care, you will remain in the hospital for about 3-4 weeks after the transplant. After you are released from the hospital, you will continue as an outpatient in the Houston area to be monitored for infections and transplant-related complications.

You will be taken off study about 100 days after the transplant. You may be taken off study early if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Azacitidine, vorinostat, gemcitabine, busulfan, melphalan, and rituximab are all FDA approved and commercially available. The use of these study drugs in combination is investigational.

Up to 60 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15 to 65 years.
2. Patients with Hodgkin's lymphoma with one or more of the following: a) Less than complete response to first-line chemotherapy. b) Relapse within 12 months of completion of first-line chemotherapy. c) Relapse within a prior irradiation field. d) Less than complete metabolic response to second-line chemotherapy. e) Second relapse or beyond. f) Extranodal disease at the time of relapse. g) Presence of B symptoms at the time of persistent disease upon completion of first-line chemotherapy, relapse or progressive disease. h) Bulky disease (defined as any lesion greater than 5 cm) at the time of persistent disease upon completion of first-line chemotherapy, relapse or progressive disease.
3. Patients with non-Hodgkin's lymphoma and one or more of the following: 1. Diffuse large B-cell lymphoma with one or more of the following: a) Primary refractory disease. b) Relapse within 12 months of completion of first-line therapy. c) Secondary IPI >1. d) Less than PR to first-line salvage chemotherapy. e) Kinetic failure after salvage chemotherapy; f) Prior treatment with 3 or more lines of therapy. g) Patients with double-hit or triple-hit NHL, in any state of the disease. 2. Peripheral T-cell lymphoma not otherwise specified (PTCL-NOS) in any stage of the disease. 3. Angioimmunoblastic T-cell lymphoma (AITL) in any stage of the disease. 4. Refractory or recurrent Burkitt¹s lymphoma. 5. Any other lymphoma that is refractory or relapsed and that does not qualify for treatment protocols of higher priority.
4. Adequate renal function, as defined by estimated serum creatinine clearance >/=50 ml/min (MDRD method from National Kidney Disease Education Program, NKDEP) and/or serum creatinine </= 1.8 mg/dL.
5. Adequate hepatic function, as defined by SGOT and/or SGPT </= 3 x upper limit of normal; serum bilirubin and alkaline phosphatase </= 2 x upper limit of normal.
6. Adequate pulmonary function with FEV1, FVC and DLCO >/= 50% of expected corrected for hemoglobin.
7. Adequate cardiac function with left ventricular ejection fraction >/= 40%. No uncontrolled arrhythmias or symptomatic cardiac disease.
8. Zubrod performance status <2.
9. Negative Beta HCG text in a woman with child-bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization.

Exclusion Criteria:

1. Patients with grade >/= 3 non-hematologic toxicity from previous therapy that has not resolved to </= grade 1.
2. Patients with prior whole brain irradiation.
3. Patients with active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA >/=10,000 copies/mL, or >/= 2,000 IU/mL).
4. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
5. Patients with active inflammatory bowel disease.
6. Active infection requiring parenteral antibiotics.
7. HIV infection, unless the patient is receiving effective antiretroviral therapy with undetectable viral load and normal CD4 counts.
8. Patients having received radiation therapy in the month prior to enrollment.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11-07 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yago Nieto, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled at MD Anderson Clinic between November 2013 and May 2015.
Groups:
- Azacitidine Dose Level 1: Azacitidine 15 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)
- Azacitidine Dose Level 2: Azacitidine 25mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)
- Azacitidine Dose Level 3: Azacitidine 35 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto Stem Cell Transplant (SCT)
Period: Overall Study
Arm/Group | Azacitidine Dose Level 1 | Azacitidine Dose Level 2 | Azacitidine Dose Level 3
Started | 37 | 19 | 5
Completed | 37 | 18 | 5
Not Completed | 0 | 1 | 0
Not completed — Disease Progression | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Azacitidine Dose Level 1: Azacitidine 15 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
- Azacitidine Dose Level 2: Azacitidine 25 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
- Azacitidine Dose Level 3: Azacitidine 35 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
- Total: Total of all reporting groups
Arm/Group | Azacitidine Dose Level 1 | Azacitidine Dose Level 2 | Azacitidine Dose Level 3 | Total
Number analyzed (Participants) | 37 | 18 | 5 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 1
  Between 18 and 65 years | 36 | 18 | 5 | 59
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 42.5 [17 to 65] | 41 [23 to 61] | 38 [19 to 58] | 41 [17 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 3 | 25
  Male | 23 | 10 | 2 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 0 | 9
  White | 20 | 9 | 4 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 3 | 1 | 16
Region of Enrollment [Number; unit: participants]
  United States | 37 | 18 | 5 | 60
Overall Study Group [Number; unit: participants]
  Disease-DLBCL | 18 | 7 | 1 | 26
  Disease-Hodgkin lymphoma | 12 | 6 | 3 | 21
  Disease-T-cell lymphoma | 5 | 3 | 0 | 8
  Disease-Other B-cell lymphoma | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Frequency of DLT
Description: Maximum tolerated dose (MTD) of azacitidine based on DLT was defined as any Grade 4 nonhematologic and noninfectious toxicity or any grade 3 mucositis or skin toxicity lasting > 3 days at peak severity. For dose finding, the continunal reassessment method was used with a target DLT probability per cohort of 25%. Azacitidine doses were chosen adaptively for sucessive cohorts with a minimum size of 2 patients. Toxicity scoring followed the National Cancer Institute Common Toxicity Criteria, version 3.
Time Frame: Enrollment up to day 30 post transplant for each dosing cohort
Measure: Number; unit: Dose-limiting toxicities
Arm/Group | Azacitidine Dose Level 1 | Azacitidine Dose Level 2 | Azacitidine Dose Level 3
Number analyzed (Participants) | 37 | 18 | 5
Dose-limiting toxicities | 16 | 28 | 40

2. Primary Outcome: Participants With Event-free Survival (EFS)
Description: EFS is defined as the time from transplantation to either relapse, second tumors, or death, whichever occurred first, or last contact. EFS was analzyed by the individual disease groups rather than the cohort dose levels.
Time Frame: Enrollment up to 100 days post transplant.
Measure: Count of Participants; unit: Participants
Groups:
- DLBCL: DLBCL patients who received the following: Azacitidine 15 mg/m2-35 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
- Hodgkin Lymphoma: Hodgkin Lymphoma patients who received the following: Azacitidine 15 mg/m2-35 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
- T-cell NHL: T-cell NHL patients who received the following: Azacitidine 15 mg/m2-35 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
- Other B-cell Lymphoma: Other B-cell lymphoma (Follicular lymphoma and Mantle cell lymphoma) who received the following: Azacitidine 15 mg/m2-35 mg/m2 IV for 10 days+Vorinostat 1000 mg PO for 10 days+ Busulfan (adjusted PK dosing) IV for 4 days+Gemcitabine 2775 mg/m2 IV for 2 days+Melphalan 60 mg/m2 IV for 2 days +/- Rituximab 375 mg/m2 IV for 1 day (for CD20 positive tumors)+ Auto SCT
Arm/Group | DLBCL | Hodgkin Lymphoma | T-cell NHL | Other B-cell Lymphoma
Number analyzed (Participants) | 26 | 21 | 8 | 5
Participants | 17 | 16 | 7 | 5

ADVERSE EVENTS:
Time Frame: Up to 100 Days post autologous transplant.
Arm/Group | Azacitidine Dose Level 1 | Azacitidine Dose Level 2 | Azacitidine Dose Level 3
All-Cause Mortality (participants affected / at risk) | 1/37 | 0/18 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/18 | 0/5
Other Adverse Events (participants affected / at risk) | 37/37 | 18/18 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azacitidine Dose Level 1 (N=37) | Azacitidine Dose Level 2 (N=18) | Azacitidine Dose Level 3 (N=5)
Hypertension (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
DVT (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Fever (General disorders) | 4 (4) | 2 (2) | 0 (0)
Fluid Overload (General disorders) | 21 (21) | 9 (9) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 26 (26) | 12 (12) | 2 (2)
Mucositis (Gastrointestinal disorders) | 34 (34) | 17 (17) | 5 (5)
Nausea (Gastrointestinal disorders) | 34 (34) | 15 (15) | 5 (5)
Elevated Creatinine (Renal and urinary disorders) | 7 (7) | 1 (1) | 2 (2)
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 24 (27) | 13 (15) | 1 (1)
Elevated Bilirubin (Hepatobiliary disorders) | 15 (15) | 9 (9) | 3 (3)
Infection (Infections and infestations) | 14 (24) | 7 (9) | 4 (4)
Neutropenic Fever (Infections and infestations) | 37 (38) | 16 (16) | 5 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 21 (21) | 6 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT01983969/Prot_SAP_000.pdf